CLINICAL TRIAL: NCT01042457
Title: Concentration-controlled Therapy of Mycophenolate Mofetil (MMF) in Proliferative Lupus Nephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-002
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Lupus Nephritis
Keywords: trough level; therapeutic drug monitoring; Mycophenolate mofetil; Mycophenolic acid; lupus nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mycophenolate mofetil (Other)
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — Drug : Mycophenolate Mofetil. Starting doses : 1000-1500 mg/day with titration based on Mycophenolic 1-hour post dose level.
  Other Names: cellcept

SUMMARY:
To evaluate therapeutic response to MMF treatment in patients with International Society of Nephrology/Renal Pathology Society (ISN/RPS) class III or IV lupus nephritis. Mycophenolic acid levels at 1-hour post dose will be monitored monthly up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-60 years.
* Ability and willingness to provide written informed consent (or to obtain consent from parent guardian where applicable) and to comply with the schedule of protocol requirements
* Diagnosis of SLE according to ACR criteria. At least 4 criteria must have been present for the diagnosis of SLE. The 4 criteria do not have to be present at the time of screening
* Active lupus nephritis defined as follows: Biopsy proven (within 16 weeks prior to screening) ISN Class III or IV (A or A/C) not include III(C) IV(C) and VI (>90% chronic irreversible scarring)

Exclusion Criteria:

Relates to SLE

* Severe renal impairment as defined by calculated creatinine clearance or MDRD-GFR < 30 ml/min(except creatinine clearance or MDRD-GFR > 50 ml/min in the 12 weeks prior to screening)
* History of serious disease or complication in any organ system that not appropriate to treatment immunosuppressive drug groups.

Related to Treatment

* Previous of any Mycophenolate groups in the 3 months prior to screening.
* Treatment with more than 2 g Cyclophosphamide in the last 6 months period prior to screening.
* Receipt of more than 3 g IV pulse methylprednisolone within the last 3 months prior to screening.
* Receipt of prednisolone dose > 30 mg/day for longer than 30 days within last 3 months prior to screening.

Related to General Health

* Pregnancy or breast feeding mothers.
* Evidence of significant uncontrolled concomitant disease in any organ system not related to SLE.
* History of cancer, including solid tumors, hematological malignancies and carcinoma.
* History of serious recurrent or chronic infection.
* Evidence of current abuse of drugs or alcohol.

Related to Laboratory Findings

* Neutrophile < 1,500/mm3, Hb < 7g/L, Platelet < 50,000/mm3 (except active SLE)
* Positive HBsAg or anti-HCV or anti-HIV.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Response rate of Mycophenolic acid concentration-controlled therapy in active lupus nephritis patients at 6th month | 24 weeks

SECONDARY OUTCOMES:
To determine Mycophenolic acid level related side effect. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yingyos Avihingsanon, MD, Study Director — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: (Lupus Research Unit) — http://www.lupus.research.chula.ac.th/